CLINICAL TRIAL: NCT02109341
Title: Phase I/II Study to Evaluate Nab-paclitaxel in Substitution of CPT11 or Oxaliplatin in FOLFIRINOX Schedule as First Line Treatment in Metastatic Pancreatic Cancer
Acronym: NabucCO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gruppo Oncologico Italiano di Ricerca Clinica (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Goirc 01-2013; 2013-002275-18 (EudraCT Number)
Record Dates: First submitted 2014-04-02; First posted 2014-04-09 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: mPC
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nab-FOLFIRI (Experimental): In the phase I study, all pts enrolled in this arm will receive Nab-FOLFIRI: Irinotecan, 180 mg per square meter of body surface area (m2 ) + Leucovorin, 400 mg/m2 and 5-Fluorouracil, 400 mg/m2 given as a bolus followed by 2400 mg/m2 given as a 46-hour continuous infusion, plus Nab-p per cohort escalation assignment starting with 90 mg/m2 every 2 weeks. Pts continued treatment until a total of 12 administrations, disease progression or unacceptable toxicity.
  Pts enrolled in arm A for phase II will receive the dose of Nab-FOLFIRI as determined in the Phase I and in the same sequence.
  Interventions: Drug: Paclitaxel bound albumine
- Nab-FOLFOX (Experimental): In the phase I study, all pts enrolled in this arm will receive Nab-FOLFOX: Oxaliplatin 85 mg/m2 +Leucovorin, 400 mg/m2 and 5-Fluorouracil, 400 mg/m2 given as a bolus followed by 2400 mg/m2 given as a 46-hour continuous infusion, plus Nab-p per cohort escalation assignment starting with 90 mg/m2, every 2 weeks.
  Pts continued treatment until a total of 12 administrations, disease progression or unacceptable toxicity.
  Pts enrolled in arm B for phase II will receive the dose of Nab-FOLFOX as determined in the Phase I and in the same sequence
  Interventions: Drug: Paclitaxel bound albumine

INTERVENTIONS:
Drug: Paclitaxel bound albumine
  Other Names: nab-paclitaxel

SUMMARY:
At this moment, FOLFIRINOX is the best treatment for selected patients (pts) with metastatic pancreatic cancer (mPC). Investigator would like to evaluate the substitution of CPT11 or Oxaliplatin in FOLFIRINOX schedule with Nab-paclitaxel (Nab-p) [Nab-FOLFIRI and Nab-FOLFOX].

Doses for Nab-FOLFIRI and Nab-FOLFOX will be determined by the phase I trial. One or both schedules will be evaluated in successive phase II part.

DETAILED DESCRIPTION:
The primary objective for phase I of the study is to determine the MTD of Nab-p when used in substitution of OXA or CPT11 in FOLFIRINOX schedule, as first-line treatment in pts with mPC. The dose finding strategy will be based on the classical 3+3 dose escalation design.

-Analysis sets: Modified intention-to-treat population: it consists of all pts who are allocated and receive at least one dose of any component of study treatment. Pts will be grouped according to the randomized treatment assignment. Pts treated during the phase I step will be not included in this population.

Safety population: it consists of all pts who are allocated and receive at least one dose of any component of study treatment. Groups are defined by the study treatment actually received. Pts treated at the MTD during the phase I step will be not included in this population.

Statistical methods Best ORR will be summarized and 95% confidence limits will be calculated according to the exact method for each of the treatment arms included in the phase II step.

All the analyses of primary and secondary efficacy variables will be performed on the modified intention-to-treat population.

The overall incidences of AEs will be summarized. Pts who experienced the same event on more than one occasion are counted only once in the calculation of the event frequency, at the highest intensity ever observed.

Serious adverse events will be summarized. All the safety analyses will be performed on the safety population.

-Sample size: The experimental treatment, to be considered clinically worthwhile, should determine an overall best RR equal to or greater than 40%. According to the Fleming single stage design, for a 90% power towards an alternative hypothesis of an ORR equal to or greater than 40% and a one-sided type I error rate of 5%, respect to the null hypothesis of an ORR equal to or less than 20%, 42 pts must be included in the final evaluation, in each arm of the phase II step. According to the exact binomial test, the experimental treatment will be considered sufficiently promising and candidate to further studies in the case of a major objective response is seen in at least 14 pts.

ELIGIBILITY:
Inclusion Criteria:

* . Males or females ≥ 18 years old and ≤ 75 years old;
* Histological or cytological evidence of a diagnosis of pancreatic ductal adenocarcinoma;
* Written informed consent prior to any study-specific procedures; 4. Measurable metastatic disease, defined in according to RECIST Version 1.1 (Eisenhower et al. 2009), that had not previously been treated with CT for metastatic disease;
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 or 1 ;
* Absence of previous abdominal radiotherapy on target lesions (except radiation therapy analgesic if it has not been performed on measurable targets);
* Absence of heart failure or angina or infarction within 12 months previous inclusion;
* Have adequate organ function including:

Hematologic: absolute neutrophil count (ANC) ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L.

Hepatic: Bilirubin ≤ 1.5 times upper limits of normal (ULN) (Pts may have endoscopic or radiologic stenting to treat biliary obstructions).

Renal: Serum creatinine within normal limits ≤1.5 times ULN.

Exclusion Criteria:

* Age of 76 years or older;
* Endocrine or acinar pancreatic carcinoma;
* Previous radiotherapy for measurable lesions;
* Central nervous system metastasis;
* Other concomitant cancer or history of cancer outside a carcinoma in situ of the cervix or basal or squamous cell of the skin;
* Pts already included in another clinical trial with other experimental drugs;
* Current active infection;
* Have serious pre-existing medical conditions or serious concomitant systemic disorders that would compromise the safety of the patient or his/her ability to complete the study, at the discretion of the investigator (for example, unstable angina pectoris, or a clinically significant history of cardiac disease or uncontrolled diabetes mellitus);
* Females who are pregnant or lactating;
* Unable to undergo medical test for geographical, social or psychological reason
* Known dihydropyrimidine dehydrogenase (DPD) deficiency

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Dose finding safety and activity | 18 months
  To determine the maximum tolerated dose (MTD) and dose-limiting toxicities (DLTs) of the combination Nab-paclitaxel+ Irinotecan+ Leucovorin+ 5-Fluorouracil (Nab-FOLFIRI) and of the combination Nab-paclitaxel+ Oxaliplatin+ Leucovorin+ 5-Fluorouracil (Nab- FOLFOX) in pts with mPC in first-line chemotherapy (CT).
  To assess efficacy of Nab-FOLFIRI and Nab-FOLFOX in pts with mPC in first-line CT , in term of ORR [Complete response (CR) + partial responses (PR)].

SECONDARY OUTCOMES:
Clinical benefit rate [CR+PR+ stable diseases (SD)] | 18 months
  - Clinical benefit rate [CR+PR+ stable diseases (SD)]: this is defined as the occurrence of either a confirmed CR or PR objective response or a SD over the entire course of treatment, as determined by the RECIST 1.1 criteria based on investigator assessment. Pts for whom no records of post-baseline tumor assessments are reported will be counted as non-responders
Progression free survival (PFS) for each schedule | 18 months
  - Duration of PFS: this is defined as the time between the date of randomization and the date of first evidence of progressive disease or date of death, whichever occurs first. Documentation of disease progression will be defined as per RECIST 1.1 criteria based on investigator assessment. The censoring date for a patient who is known to be progression-free would be the date of the last tumor assessment.
Overall survival (OS), | 18 months
  - Duration of OS: is the time from the date of randomization to the date of death from any cause. For pts who are still alive on the date of clinical data cut-off for the OS analysis, the last date when the patient is known to be alive on or prior to the clinical cut-off date will be used to determine the censoring date. For pts who do not have any post-baseline information, data will be censored at the date of randomization plus one day.
Quality of life (QoL) for each schedule | 18 months
  - QoL : assessment of quality of life with the use of the European Organization for Research and Treatment of Cancer (EORTC) quality-of-life core questionnaire (QLQ-C30, version 3.0). The primary QoL endpoint will be the time to a definitive 5% deterioration in the global health status/QoL scale of the QLQ-C30 questionnaire.
Safety profile | 18 months
  - Safety profile: Safety of the treatment will be evaluated by serious and non serious adverse events (AEs). AEs will be graded according to the CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Di Costanzo, MD, Principal Investigator — AOU- Careggi; Elisa Giommoni, MD, Principal Investigator — Gruppo Oncologico Italiano di Ricerca Clinica
Locations (8):
- Italy (8):
  - Ospedale Sacro cuore di Gesù - FATEBENEFRATELLI, Benevento, BN
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, FG
  - SC Oncologia Medica 1, Florence, FI
  - Regina Elena National Cancer Institute, Rome, Rome
  - Azienda Ospedaliera Istituti Ospedalieri di Cremona, Cremona
  - Ospedale S. Chiara - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Ospedale Borgo Roma, Verona

REFERENCES:
- See also: Goirc Web site — http://www.goirc.org/